CLINICAL TRIAL: NCT05507918
Title: Effect of Pre-operative Oral Hydration on Post-operative Pain and Nausea in Adults Undergoing Tonsillectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: limitations in staff and resources
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Matthew Farrugia, Program Director, Otolaryngology Head and Neck Residency Program, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-017
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Tonsil Disease; Surgical Wound; Pain, Postoperative
Keywords: Oral hydration; Tonsillectomy; Adult Surgery; Pain Control
MeSH Terms: conditions — Surgical Wound; Pain, Postoperative; Agnosia | interventions — Water

STUDY DESIGN:
Intervention Model Description: 3 group parallel comparison, non-blinded, interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low fluid intake (Experimental): 0.5 L - 1.5 L fluid intake in the 24 hours prior to NPO status for surgery
  Interventions: Other: Oral water and clear liquids
- Medium fluid intake (Experimental): 1.5 L - 3 L fluid intake in the 24 hours prior to NPO status for surgery
  Interventions: Other: Oral water and clear liquids
- High fluid intake (Experimental): 3 L - 4.5 L fluid intake in the 24 hours prior to NPO status for surgery
  Interventions: Other: Oral water and clear liquids

INTERVENTIONS:
Other: Oral water and clear liquids — Measured oral intake of fluids prior to tonsillectomy
  Other Names: Oral Hydration

SUMMARY:
Tonsillectomy is commonly described as one of the most painful procedures that an adult can undergo. This study's aim is to evaluate if pre-operative oral hydration has an impact in reducing post-operative pain, nausea and vomiting, and opioid medication use after adult tonsillectomies. Participants will be randomized to a low, medium and high fluid intake groups and will record fluid intake on the day before surgery. After surgery, participants will record their pain and nausea at timepoints up to 7 days post-operative. Medication use will be recorded up to the first post-operative follow-up visit with their physician.

DETAILED DESCRIPTION:
Common indications for adult tonsillectomy include tonsillar hypertrophy, obstructive sleep apnea, and chronic tonsillitis. Although there are many studies looking into how best to prevent and treat post-operative pain and nausea, there are very few that give recommendations to the patients pre-operatively. This study's aim is to evaluate if pre-operative oral hydration has an impact in reducing post-operative pain, nausea and vomiting after adult tonsillectomies. If pre-operative hydration can reduce the pain associated with the procedure, then this could also be an adjunct to help reduce the amount of narcotic pain medication that is required.

The goal of this study is to evaluate if the amount of pre-operative oral hydration can reduce the amount of pain and nausea/vomiting in patients undergoing adult tonsillectomies. This study will be measuring post-operative pain and nausea scores at several points after the adult tonsillectomy procedure for participants that have consumed different amounts of clear fluid in the 24 hours leading up to their nothing by mouth (NPO) status. Participants will be randomized to one of three categories of preoperative fluid: 0.5 - 1.5 Liters (L), 1.5 - 3 L, and 3 - 4.5 L, which will correlate to the low, medium and high fluid intake groups, respectively. Participants will be given a 1000 mL measuring water bottle that they can use to accurately record their fluid consumption in the 24 hours prior to their pre-operative NPO status. The fluid consumption that they record will include all liquids (i.e., water, flavored water, juice, coffee, tea, soda, milk, alcohol). They will be asked to keep a record of the volume of caffeinated beverage versus un-caffeinated beverages.

After surgery the participants will be given a form to record their pain and nausea scores. Participants will record their pain and nausea by using two separate 10-point scales at 7 different points after the procedure. These scores will be measured immediately after surgery, and at 4 hours, 8 hours, 24 hours, 72 hours, 5 days and 7 days postoperative. This form, along with a count of opioid medication used, will be retuned to the physician at the first post-operative follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult undergoing primary tonsillectomy or any procedure which includes tonsillectomy as component at Beaumont Farmington Hills Hospital or Novi Surgery Center.
* Patients greater than or equal to 18 years of age

Exclusion Criteria:

* Patients < 18 years of age
* Decisionally impaired
* Adults with history of significant gastro-esophageal pathology (ie. gastric/duodenal ulcers, Barrett's esophagus, eosinophilic esophagitis)
* Patient undergoing tonsillectomy procedure due to previous or active peri-tonsillar abscess or for resection of cancer
* Allergy or contraindication to the use of acetaminophen or narcotic medications
* Pregnant
* Patients that have chronic disease states including chronic kidney disease, congestive heart failure, diabetes mellitus, diabetes insipidus, or chronic pain syndrome
* Patients that are on chronic pain medications, diuretics or steroids
* Patients that have history of significant nausea/vomiting associated with anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pain 8 hours postoperative | 8 hours postoperative
  Participant reported pain on a Likert scale from 0-10, where 0=no pain and 10= worst pain possible.
Nausea 4 hours postoperative | 4 hours postoperative
  Participant reported nausea on a Likert scale from 0-10, where 0=no nausea and 10 = worst nausea possible.

SECONDARY OUTCOMES:
Pain postoperative | up to 7 days postoperative
  Participant reported pain on a Likert scale from 0-10, where 0=no pain and 10= worst pain possible.
Nausea postoperative | up to 7 days postoperative
  Participant reported nausea on a Likert scale from 0-10, where 0=no nausea and 10 =
Narcotic pain medication use immediately following surgery | 4 hours
  Opioid pain medication administered in Post-Anesthesia Care Unit (PACU) in morphine equivalents
Nausea medication use immediately following surgery | 4 hours
  Oral anti-nausea medication administered in Post-Anesthesia Care Unit (PACU)
Narcotic pain medication use after discharge | up to 14 days postoperative
  Opioid pain medication used after discharge in morphine equivalents
Nausea medication use after discharge | up to 14 days postoperative
  Oral anti-nausea medication (4 mg zofran) used after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Farrugia, DO, Principal Investigator — Beaumont Health - Farmington Hills

IPD SHARING:
Plan to Share IPD: No